CLINICAL TRIAL: NCT03554746
Title: Additional Gluteal Control Training for Low Back Pain With Functional Leg Length Inequality: A Ramdomized Controlled Trail
Brief Title: Additional Gluteal Control Training for Low Back Pain With Functional Leg Length Inequality
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Yang Ming Chiao Tung University (Other)
Responsible Party: Principal Investigator, Yi-Fen Shih, Professor, Department of Physical Therapy and Assistive Technology, National Yang-Ming University, National Yang Ming Chiao Tung University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: YM106055F
Record Dates: First submitted 2018-05-30; First posted 2018-06-13 (Actual); Results first posted 2019-09-19 (Actual); Last update posted 2019-09-19 (Actual); Status verified 2019-08

CONDITIONS: Low Back Pain, Recurrent
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GC group (Experimental): It mainly involve core stability exercise, stretching exercise and gluteal control training. All of above will be arranged 3 times a week for a total 6 weeks.
  Interventions: Other: GC group
- CG group (Experimental): It involve core stability exercise and stretching exercise. All of above will be arranged 3 times a week for a total 6 weeks.
  Interventions: Other: CG group

INTERVENTIONS:
Other: GC group — 1. core stability training: hold 5s/rep, 20 reps/times
     1. supine, pelvic posterior tilt with TrA contraction.
     2. supine, pelvic posterior tilt and maintain bil. knee on 90 degrees.
     3. All four position with leg raise
  2. Stretching ex. : hold 15 s/reps, 5 reps/times
     1. Hamstring
     2. Quadriceps
  3. Additional gluteal muscle control training: hold 10 s/reps, 20 reps/times 1st to 2nd:
     1. clam ex. without resistance
     2. single leg bridge with maintain bil. ASIS even level 3rd to 4th: maintain 1st to 2nd ex. with resistance 5th:
     <!-- -->
     1. maintain 3rd to 4th ex.
     2. single leg standing on rock board to maintain balance 6th:
     <!-- -->
     1. maintain 5th ex.
     2. lunge ex. without hip internal rotation
  Other Names: Additional gluteal muscle control training
  Arms: GC group
Other: CG group — 1. core stability training: hold 5s/rep, 20 reps/times
     1. supine, pelvic posterior tilt with TrA contraction.
     2. supine, pelvic posterior tilt and maintain bil. knee on 90 degrees.
     3. All four position with leg raise
  2. Stretching ex. : hold 15 s/reps, 5 reps/times
     1. Hamstring
     2. Quadriceps
  Other Names: General core strengthening
  Arms: CG group

SUMMARY:
Low back pain (LBP) is a prevalent musculoskeletal disorder. A variety of exercise interventions which were designed as randomized control trails (RCTs) have been studied and shown effectiveness in improving pain and disability. These exercises typically focus on the abdominal and back musculature strength. However, many LBP patients did not show any improvement in their symptom after they carry out those exercise programs.

DETAILED DESCRIPTION:
Low back pain (LBP) is a prevalent musculoskeletal disorder. A variety of exercise interventions which were designed as randomized control trails (RCTs) have been studied and shown effectiveness in improving pain and disability. These exercises typically focus on the abdominal and back musculature strength. However, many LBP patients did not show any improvement in their symptom after they carry out those exercise programs. Some authors consider that this type of low back pain may be caused by leg length inequality (LLI) in these patients, which resulted from poor gluteal neuromuscular control or muscles' imbalance.

In consideration of few studies have been done for investigating the effects of gluteal muscles control training in LBP. Thus, the purpose of this study is to investigate the effect of additional gluteal muscles control training on improving functional LLI in patients with LBP. We hypothesized that gluteal muscle control training would be more effective in self-reported pain, and their functional disability would be improve after 6-week training program than control training group.

ELIGIBILITY:
Inclusion Criteria:

* non-specific LBP (from inferior rib margin to the gluteal fold)
* more than 3 months
* Visual Analog Scale ≧5 (in past one month)
* pelvic innominate rotation (anterior rotation in dominant side)

Exclusion Criteria:

* history of fracture or surgery
* congenital anomalies in the spine, pelvis, or lower limbs
* recent trauma, tumor, pregnancy or scoliosis
* lower extremity paresthesia, unknown weakness
* bowel and bladder dysfunction
* predominant lower extremity pain with standing
* presence of system illness, no reasoning weight loss, predominant night pain
* specific sacroiliac joint dysfunction

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2017-12-11 (Actual); Primary Completion 2018-07-23 (Actual); Study Completion 2018-09-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yi-Fen Shih, PhD, Study Director — Department of Physical Therapy and Assistive Technology, National Yang-Ming University
Locations (1):
- National Yang Ming University, Taipei, Taiwan

RESULTS

PARTICIPANT FLOW:
Groups:
- GC Group: It mainly involve core stability exercise, stretching exercise and gluteal control training. All of above will be arranged 3 times a week for a total 6 weeks.
  GC group: 1. core stability training: hold 5s/rep, 20 reps/times supine, pelvic posterior tilt with TrA contraction. supine, pelvic posterior tilt and maintain bil. knee on 90 degrees. All four position with leg raise 2. Stretching ex. : hold 15 s/reps, 5 reps/times
  a. Hamstring b. Quadriceps 3. Additional gluteal muscle control training: hold 10 s/reps, 20 reps/times
  1st to 2nd: clam ex. without resistance single leg bridge with maintain bil. ASIS even level 3rd to 4th: maintain 1st to 2nd ex. with resistance 5th:
  a. maintain 3rd to 4th ex. b. single leg standing on rock board to maintain balance 6th: maintain 5th ex. lunge ex. without hip internal rotation
- CG Group: It involve core stability exercise and stretching exercise. All of above will be arranged 3 times a week for a total 6 weeks.
  CG group: 1. core stability training: hold 5s/rep, 20 reps/times supine, pelvic posterior tilt with TrA contraction. supine, pelvic posterior tilt and maintain bil. knee on 90 degrees. All four position with leg raise 2. Stretching ex. : hold 15 s/reps, 5 reps/times
  a. Hamstring b. Quadriceps
Period: Overall Study
Arm/Group | GC Group | CG Group
Started | 24 | 24
Completed | 24 | 24
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- CG Group: IIt involve core stability exercise and stretching exercise. All of above will be arranged 3 times a week for a total 6 weeks.
  CG group: 1. core stability training: hold 5s/rep, 20 reps/times supine, pelvic posterior tilt with TrA contraction. supine, pelvic posterior tilt and maintain bil. knee on 90 degrees. All four position with leg raise 2. Stretching ex. : hold 15 s/reps, 5 reps/times
  a. Hamstring b. Quadriceps
- Total: Total of all reporting groups
Arm/Group | GC Group | CG Group | Total
Number analyzed (Participants) | 24 | 24 | 48
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.58 (9.42) | 47.38 (11.31) | 47.48 (10.47)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 14 | 27
  Male | 11 | 10 | 21
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Leg Length Inequality
Description: functional leg length inequality
Time Frame: change from baseline at 6 weeks later
Measure: Mean (Standard Deviation); unit: centemeter
Groups:
- GC Group: It mainly involve core stability exercise, stretching exercise and gluteal control training. All of above will be arranged 3 times a week for a total 6 weeks.
  GC group: 1. core stability training: hold 5s/rep, 20 reps/times
  1. supine, pelvic posterior tilt with TrA contraction.
  2. supine, pelvic posterior tilt and maintain bil. knee on 90 degrees.
  3. All four position with leg raise 2. Stretching ex. : hold 15 s/reps, 5 reps/times
  a. Hamstring b. Quadriceps 3. Additional gluteal muscle control training: hold 10 s/reps, 20 reps/times
  1st to 2nd:
  1. clam ex. without resistance
  2. single leg bridge with maintain bil. ASIS even level 3rd to 4th: maintain 1st to 2nd ex. with resistance 5th:
  a. maintain 3rd to 4th ex. b. single leg standing on rock board to maintain balance 6th:
  1. maintain 5th ex.
  2. lunge ex. without hip internal rotation
- CG Group: It involve core stability exercise and stretching exercise. All of above will be arranged 3 times a week for a total 6 weeks.
  CG group: 1. core stability training: hold 5s/rep, 20 reps/times
  1. supine, pelvic posterior tilt with TrA contraction.
  2. supine, pelvic posterior tilt and maintain bil. knee on 90 degrees.
  3. All four position with leg raise 2. Stretching ex. : hold 15 s/reps, 5 reps/times
  a. Hamstring b. Quadriceps
Arm/Group | GC Group | CG Group
Number analyzed (Participants) | 24 | 24
centemeter | 0.3 (0.21) | 0.58 (0.13)

2. Primary Outcome: Ilium Anterior Tilt Difference
Description: bilateral ilium anterior tilt difference
Time Frame: change from baseline at 6 weeks later
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | GC Group | CG Group
Number analyzed (Participants) | 24 | 24
degrees | 0.67 (0.65) | 2.27 (0.65)

3. Primary Outcome: Pelvic Inclination
Description: bilateral pelvic inclination
Time Frame: change from baseline at 6 weeks later
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | GC Group | CG Group
Number analyzed (Participants) | 24 | 24
degrees | 1.03 (0.37) | 1.56 (0.51)

4. Secondary Outcome: Pain Intensity
Description: Visual Analog Scale (VAS) (0-10) Maximum: 10 Minimal: 0 higher scores mean a worse outcome
Time Frame: change from baseline at 6 weeks later
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | GC Group | CG Group
Number analyzed (Participants) | 24 | 24
score on a scale | 1.3 (1.21) | 3.44 (1.06)

5. Secondary Outcome: Functional Disability
Description: Oswestry disability index (ODI) Maximum: 100 Minimal: 0 higher scores mean a worse outcome
Time Frame: change from baseline at 6 weeks later
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | GC Group | CG Group
Number analyzed (Participants) | 24 | 24
score on a scale | 7.51 (5.34) | 11.91 (6.65)

6. Secondary Outcome: Functional Ability
Description: PSFS (0-10) Maximum: 10 Minimal: 0 higher scores mean a better outcome
Time Frame: change from baseline at 6 weeks later
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | GC Group | CG Group
Number analyzed (Participants) | 24 | 24
score on a scale | 8.23 (1.18) | 7.09 (1.28)

ADVERSE EVENTS:
Time Frame: The time frame is 9 months (Study Start Date: December 11, 2017 to the Study Completion Date: September 10, 2018). After all the included participants complete the intervention and pre/post tests.
Description: Results submission is required by FDAAA 801 for certain applicable clinical trials of drugs, biologics and devices.
  This study was an exercise intervention for low back pain patients. We didn't use any drugs, biologics and devices.
Arm/Group | CG Group | GC Group
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/24
Other Adverse Events (participants affected / at risk) | 0/24 | 0/24

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-05-30): https://cdn.clinicaltrials.gov/large-docs/46/NCT03554746/Prot_SAP_000.pdf